CLINICAL TRIAL: NCT05022667
Title: Assessing Benefits of Near Infrared Autofluorescence (NIRAF) Detection for Identifying Parathyroid Glands During Total Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Paul Gauger, Ambulatory Care Clinical Chief, William J Fry Professor of Surgery and Professor of Surgery, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00194322
Record Dates: First submitted 2021-08-22; First posted 2021-08-26 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Neoplasms; Thyroid Diseases; Hypoparathyroidism; Endocrine System Diseases; Endocrine Gland Neoplasms; Neoplasms by Site; Neoplasms; Head and Neck Neoplasms; Parathyroid Diseases
Keywords: Total Thyroidectomy; Intraoperative Parathyroid Identification; Near Infrared Autofluorescence; Postoperative Hypocalcemia; Postoperative Hypoparathyroidism
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases; Hypoparathyroidism; Endocrine System Diseases; Endocrine Gland Neoplasms; Neoplasms by Site; Neoplasms; Head and Neck Neoplasms; Parathyroid Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PTeye (Experimental): The surgeon will use the PTeye as an intraoperative tool to identify if a suspect tissue is a parathyroid or not, during the total thyroidectomy procedure.
  Interventions: Device: PTeye
- Standard of Care (No Intervention): The surgeon will not use the PTeye and will proceed with the total thyroidectomy as usual, while relying solely on her/his surgical experience in identifying the parathyroid glands during the operations.

INTERVENTIONS:
Device: PTeye — The surgeon will first take 5 baseline NIRAF measurements on the thyroid gland (or neck muscle, if thyroid is absent) using the disposable sterile fiber probe that is connected to the PTeye console, as per device functionality requirements.
  Arms: PTeye

SUMMARY:
This study will see if the use of near infrared autofluorescence (NIRAF) detection with a 'Parathyroid Eye (PTeye)' for identifying parathyroid glands (PGs) during total thyroidectomy (TTx) is better than surgeon's detection alone. It compares risk, benefits and outcomes in TTx patients where NIRAF detection with PTeye for parathyroid identification is either used or not used.

DETAILED DESCRIPTION:
Prior to data collection, it was determined some additional outcome measures collected by the primary site would not be relevant to the trial for participating sites such as this site. Those outcomes were removed from this record.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thyroid disease who will be undergoing total thyroidectomy (includes patients who have undergone a prior neck exploration for parathyroid disease or other but have an intact thyroid gland).
* Patients with persisting thyroid disease and will be undergoing re-operative or completion thyroidectomy.

Exclusion Criteria:

* Pregnant women
* Patients with concurrent parathyroid and thyroid disease
* Patients with incidental enlarged parathyroid discovered during thyroidectomy procedure.
* Patients undergoing thyroid lobectomy or partial thyroidectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gauger, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cousart AG, Kiernan CM, Willmon PA, Thomas G, Wang TS, Gauger PG, Duh QY, Underwood HJ, Jackson A, Patel A, Mahadevan-Jansen A, Solorzano CC. Near-Infrared Autofluorescence for Parathyroid Detection During Endocrine Neck Surgery: A Randomized Clinical Trial. JAMA Surg. 2025 Sep 1;160(9):936-944. doi: 10.1001/jamasurg.2025.2233. PMID 40668552

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PTeye | Standard of Care
Started | 57 | 57
Completed (Participants were considered to have completed the trial if data was collected from them for the primary outcome measure.) | 57 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTeye | Standard of Care | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (16.9) | 52.6 (16) | 51.9 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 43 | 87
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 54 | 55 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47 | 49 | 96
  Black | 4 | 3 | 7
  Asian | 3 | 4 | 7
  Other | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 57 | 114
Preoperative calcium (pg/dL) [Mean (Standard Deviation); unit: (pg/dL)] | 9.4 (0.5) | 9.5 (0.4) | 9.5 (0.5)
Preoperative PTH (pg/mL) [Mean (Standard Deviation); unit: (pg/mL)] | 48.2 (22.4) | 78.3 (25) | 64.6 (27.9)
Preoperative vitamin D (mcg) [Mean (Standard Deviation); unit: mcg] | 33 (13.6) | 29.3 (11) | 30.9 (12)
Final Diagnosis [Count of Participants; unit: Participants]
  Grave's disease | 18 | 15 | 33
  Goiters and nodular diseases | 13 | 6 | 19
  Thyroid cancer | 26 | 36 | 62

OUTCOME MEASURES:

1. Primary Outcome: The Average Number of Parathyroid Glands Identified (Experimental Group: Glands Identified With Naked Eye + NIRAF; Control Group: Glands Identified With Naked Eye) Per Patient
Description: Overall number of parathyroid glands identified (Experimental Group: Glands identified with naked eye + NIRAF; Control Group: Glands identified with naked eye)
Time Frame: Immediate (During total thyroidectomy procedure)
Measure: Mean (95% Confidence Interval); unit: parathyroid glands per patient
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 57 | 57
parathyroid glands per patient | 3.1 [2.8 to 3.3] | 2.9 [2.6 to 3.2]
Statistical Analysis 1: Comparison: PTeye vs Standard of Care; Test type: Superiority; p = 0.3, t-test, 2 sided

2. Secondary Outcome: Blood Parathyroid Hormone (PTH) Levels at 5-14 Days After Surgery
Description: Blood parathyroid hormone (PTH) levels at 5-14 days post-op
Time Frame: 5-14 days after surgery
Population: Not all participants returned for this lab assessment during the 5-14 day data collection period. As such, no data for these participants was collected.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 35 | 36
pg/mL | 35.6 (25.3) | 41 (34.7)
Statistical Analysis 1: Comparison: PTeye vs Standard of Care; Test type: Superiority; p = .5, t-test, 2 sided

3. Secondary Outcome: Blood Parathyroid Hormone (PTH) Levels at 24-48 Hours After Surgery
Description: Blood parathyroid hormone (PTH) levels at 24-48 hours after surgery
Time Frame: Within 24-48 hours after surgery
Population: Not all participants returned for this lab assessment during the 24-48 hour data collection period. As such, no data for these participants was collected.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 56 | 52
pg/mL | 20.7 (11.6) | 24.3 (16.6)
Statistical Analysis 1: Comparison: PTeye vs Standard of Care; Test type: Superiority; p = .2, t-test, 2 sided

4. Secondary Outcome: Blood Calcium Levels 24-48 Hours After Surgery
Description: Blood calcium levels 24-48 hours after surgery
Time Frame: Within 24-48 hours after surgery
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/dL
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 54 | 52
pg/dL | 9.4 (.5) | 9.3 (.5)
Statistical Analysis 1: Comparison: PTeye vs Standard of Care; Test type: Superiority; p = 0.3, t-test, 2 sided

5. Secondary Outcome: Duration in Minutes of Surgery
Description: Duration of surgery (minutes)
Time Frame: Collected immediately following surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 57 | 57
minutes | 126.2 (39.6) | 120.3 (34.7)
Statistical Analysis 1: Comparison: PTeye vs Standard of Care; Test type: Superiority; p = .4, t-test, 2 sided

6. Secondary Outcome: Number of Frozen Section Analysis Performed.
Description: Number of frozen section analysis performed. Samples of a suspected piece of parathyroid tissue were removed and analyzed to confirm whether they were actually parathyroid tissue. Results reflect the participants who were determined to have had a frozen section conducted.
Time Frame: Collected immediately following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 57 | 57
Participants
  0 | 55 | 55
  1 or more | 2 | 2

7. Secondary Outcome: Number of Auto-transplanted Parathyroid Glands
Description: Number of auto-transplanted parathyroid glands if the parathyroid gland was accidentally excised/devascularized.
Time Frame: Immediate. During total thyroidectomy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 57 | 57
Participants
  0 | 41 | 46
  1 | 16 | 10
  2 or more | 0 | 1
Statistical Analysis 1: Comparison: PTeye vs Standard of Care; Test type: Superiority; p = .3, Chi-squared

8. Secondary Outcome: Number of Nights Spent in the Hospital After Total Thyroidectomy
Description: Number of nights spent for postoperative recovery in the hospital after the surgical procedure.
Time Frame: 0 - 4 nights after total thyroidectomy
Measure: Count of Participants; unit: Participants
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 57 | 57
Participants
  0 nights | 0 | 0
  1 night | 57 | 57
  > 1 night | 0 | 0

9. Secondary Outcome: Number of Inadvertently Resected Parathyroid Glands
Description: Number of inadvertently resected parathyroid glands when parathyroid tissue is found in the resected thyroid specimens. Results reflect the participants who had an inadvertently resected parathyroid gland.
Time Frame: Immediate (intraoperative) to 7-10 days after total thyroidectomy (as presented in the pathology report)
Measure: Count of Participants; unit: Participants
Arm/Group | PTeye | Standard of Care
Number analyzed (Participants) | 57 | 57
Participants | 5 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 6-months after surgery.
Arm/Group | PTeye | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 0/57 | 0/57

LIMITATIONS AND CAVEATS:
The median follow-up time of participants was 5-14 days post-operation. Therefore, we lack long-term follow-up (> 6 months) for the majority of the participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT05022667/Prot_SAP_000.pdf